CLINICAL TRIAL: NCT06634433
Title: Training of Trainers Program in Interprofessional Education for Health Professionals
Brief Title: Training of Trainers Program in IPE for Health Professionals
Acronym: TTP_IPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aysel Başer, Asistant Profesor, Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/97; 1129B372300447 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2024-10-06; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Training Effectiveness; Training; Education; Interprofessional Education
Keywords: Training of Trainers; Interprofessional Education; Competencies of Health Professionals; Trainer Development Program
MeSH Terms: interventions — Attitude of Health Personnel

STUDY DESIGN:
Intervention Model Description: This study employs a two-phase Training of Trainers Program (TTP) designed for health professionals. The first phase is a three-day online theoretical training, while the second phase consists of two days of face-to-face practical training. Participants were assigned to different small groups to engage in interprofessional education (IPE) activities and scenarios, facilitated by experts from various healthcare professions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training of Trainers (ToT) Program Group (Experimental): Participants in this group will receive a two-phase Training of Trainers Program (TTP) aimed at improving their skills in interprofessional education. The first phase includes three days of online theoretical training covering topics such as interprofessional communication, teamwork, and scenario-based learning. The second phase consists of two days of face-to-face practical sessions, where participants will engage in scenario-based group work and role-playing activities to reinforce skills in collaborative healthcare practices. To evaluate the effectiveness of the training program, all participants will complete a pre-test before the training and a post-test after the training
  Interventions: Behavioral: Health Personnel Attitude

INTERVENTIONS:
Behavioral: Health Personnel Attitude — The intervention consists of a two-phase Training of Trainers Program (TTP) designed for health professionals aimed at enhancing interprofessional education (IPE) skills. Phase 1 includes three days of online theoretical training, focusing on topics such as interprofessional collaboration, communication, and conflict resolution. Phase 2 involves two days of face-to-face practical sessions, where participants engage in scenario-based learning and small group discussions to apply IPE concepts. The effectiveness of the program is assessed through pre-test and post-test evaluations, measuring changes in participants' knowledge, attitudes, and competencies in interprofessional education.

SUMMARY:
This study aims to develop a training program for academicians and clinicians who educate health professionals. The program focuses on enhancing the knowledge, skills, and attitudes needed for interprofessional education and collaborative practice. The Training of Trainers Program (TTP) was conducted between February 20 and 24, 2024, and consisted of two phases: three days of online interactive theoretical training followed by two days of face-to-face practical training. The practical training included scenario-based group activities designed to develop professional skills in a collaborative environment. Participants were assessed using multiple tools, including demographic data forms, reflection and group assignments, and multiple-choice questions. Results showed that the TTP significantly improved competencies in areas such as teamwork, communication, leadership, ethics, and patient care. The program also received high satisfaction ratings from participants, highlighting the quality of the enrollment process, training content, and overall program effectiveness.

DETAILED DESCRIPTION:
Study Design Summary:

This study utilized a quasi-experimental design conducted between June 2023 and March 2024, following the principles of the Declaration of Helsinki. Ethical approval was obtained from the İzmir Democracy University Non-Interventional Ethics Committee (Approval No. 2023/97). The study was supported by TÜBİTAK under program 2237_A with project number 1129B372300447.

Training Program Design and Implementation: The Training of Trainers Program (TTP) in Interprofessional Education (IPE) was developed based on a literature review and the ADDIE instructional design model. The program spanned 40 hours, including 24 hours of synchronous online learning and 16 hours of face-to-face applied sessions. Facilitators from various universities and professions (including doctors, nurses, and other health professionals) led the training.

The first phase involved three days of online theoretical education focusing on key topics such as IPE competencies, communication, mentoring, and scenario writing. Interactive methods like surveys, gamification, and active learning platforms were used. The second phase consisted of two days of practical face-to-face training with small group work and scenario-based activities to foster interprofessional collaboration and communication.

Evaluation Methods: Participants were evaluated using a sociodemographic form, multiple-choice questions, and an IPE Competency Assessment Form (IPE-CAF) with 31 items assessing roles, teamwork, communication, leadership, ethics, and patient relationships. A Training Satisfaction Form with 17 items was also used to gather feedback. Quantitative data were analyzed using SPSS software, with statistical tests like the Wilcoxon signed-rank test and Cronbach's alpha for reliability. Qualitative data from open-ended questions were analyzed using descriptive content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Health Professionals: People working in the fields of health sciences such as medicine, dentistry, nursing, nutrition and dietetics, physiotherapy and rehabilitation, or working in academic positions in these fields.
* Trainer Experience: People who have taken part in trainings for health professionals or who will provide training.
* Collaborative Education Experience: Trainers who have previously been involved in interprofessional education processes or who plan to work in this field.
* Volunteerism: Participants who volunteered to participate in the training programme and provided the necessary permissions.
* In addition to all criteria, trainers over the age of 18

Exclusion Criteria:

* Non-Health Professionals: Those working or studying outside of medicine or health sciences will not be included in this programme.
* Those who do not meet the Participation Requirements: Those who cannot attend at least 80% of the online theoretical and face-to-face practical trainings of the programme.
* Non-Volunteers: Those who do not volunteer for the programme and individuals under the age of 18 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Improvement in Interprofessional Education Competencies | Pre-test conducted before the intervention and post-test conducted immediately after the completion of the intervention. (20-24 February))
  The primary outcome measure is the improvement in participants' competencies in interprofessional education (IPE), as assessed through pre- and post-training evaluations. Competencies include roles and responsibilities, team and teamwork, interprofessional communication, collaborative leadership, relationships with patients, recognizing patient needs, lifelong learning, and ethics. This will be measured using the IPE Competency Assessment Form (IPE-CAF), which is based on a Likert scale. Scores will be compared before and after the Training of Trainers Program to assess the effectiveness of the intervention.

SECONDARY OUTCOMES:
Training Program Satisfaction | Immediately after the completion of the TTP.
  Participants' overall satisfaction with the training program will be evaluated using the Training Satisfaction Form. This form collects feedback on areas such as the enrollment process, training content, trainer effectiveness, and overall program satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Baser, Asist. Prof., Study Director — Izmir Democracy University
Locations (1):
- İzmir Democracy University, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study is currently in the manuscript writing phase. After the data is published, it will be shared with any researchers who request it and provide a valid justification for its use.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This study is currently in the manuscript writing phase. After the data is published, it will be shared with any researchers who request it and provide a valid justification for its use within a 5-year period following publication.
Access Criteria: Researchers with a valid scientific purpose and justification will be able to request access to the individual participant data (IPD) and supporting information. Access will be granted after publication of the study results, and the data will be shared through a secure data-sharing platform upon approval of the request. All requests will be reviewed by the study team, and data will only be provided for research that aligns with the ethical guidelines of the study.